CLINICAL TRIAL: NCT06962852
Title: A Clinical Trial to Evaluate the Long-term Safety and Durability of Efficacy of BI 3720931, an Inhaled Lentiviral Vector Gene Therapy, After Single Dose Administration in a Previous Clinical Trial, in People With Cystic Fibrosis Rolled-over From a Previous Clinical Trial With BI 3720931 (Lenticlair™-ON)
Brief Title: A Long-term Study to Monitor the Health Status of People With Cystic Fibrosis Who Took Part in a Previous Study With BI 3720931 (Lenticlair™-ON)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1504-0003; 2023-504909-37-00 (Registry Identifier: CTIS); U1111-1291-2932 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: The trial is intended to assess 2 different objectives: long-term safety over 15 years and durability of efficacy over at least 2 years of BI 3720931 after single dose administration in a previous clinical trial in trial participants with cystic fibrosis (CF).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All trial participants (Experimental): All trial participants who have received at least one dose of BI 3720931 or matching placebo in a previous trial with BI 3720931.
  Trial participants who received placebo in the previous trial do not need to be followed for 15 years; once the treatment in the previous trial has been unblinded, their participation in this trial is then terminated.
  Interventions: Genetic: BI 3720931

INTERVENTIONS:
Genetic: BI 3720931 — BI 3720931

SUMMARY:
This study is for people with cystic fibrosis who took part in a previous study with a medicine called BI 3720931. The main purpose of this study is to monitor the long-term health of participants who were treated with BI 3720931 in the previous study. Participants in this study do not receive additional treatment with BI 3720931.

Participants who previously took BI 3720931 are in this study for 15 years. Participants who previously took placebo are in the study only until it is disclosed that they were in the placebo group, after which they stop. Participants who previously took BI 3720931 visit the study site about 20 times. Participants visit once every 3 months during the first 2 years.

After that, they visit once a year. During study visits, doctors check the health of the participants and note any health problems that could have been caused by BI 3720931. They also do lung function tests to see if BI 3720931 helps people with cystic fibrosis in the long term.

ELIGIBILITY:
Inclusion criteria:

1. Trial participants who participated in a previous BI sponsored trial with BI 3720931 and have received any dose of BI 3720931, or matching placebo
2. Signed and dated written informed consent in accordance with International Council for Harmonisation (ICH)-Good Clinical Practice (GCP) and local legislation prior to admission to the trial

There are no exclusion criteria for enrolment into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2048-11-24 (Estimated); Study Completion 2048-11-24 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent delayed adverse events (AEs) | up to 15 years
  Treatment-emergent delayed AEs are defined as new malignancies, new serious neurologic disorders, new serious rheumatologic or autoimmune disorders, new serious hematologic disorders, or new serious potentially product-related infections, until 15 years from enrolment

SECONDARY OUTCOMES:
Time to loss of efficacy defined as the drop to below 5% (absolute) above baseline in forced expiratory volume in 1 second, percent of predicted value (FEV1pp) | up to 15 years
Time to first pulmonary exacerbation (PEX) from last dosing | up to 15 years
Occurrence of AEs up to 2 years after enrolment | up to 2 years
Occurrence of serious adverse events (SAEs) throughout the study | up to 15 years
Occurrence of replication-competent lentivirus (RCL) throughout the study | up to 15 years

CONTACTS AND LOCATIONS:
Locations (10):
- France (2):
  - HOP Gui de Chauliac, Montpellier
  - HOP Necker, Paris
- Italy (2):
  - Istituto G. Gaslini, Genova
  - Osp. Pediatrico Bambin Gesù, Roma
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Universitari Vall D Hebron, Barcelona, Spain
- United Kingdom (4):
  - University Hospital Llandough, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com